CLINICAL TRIAL: NCT03474510
Title: Effective Pain Management During Shoulder Replacement Surgery With Either Continuous Ropivacaine Interscalene Nerve Block or Local Infiltration With EXPAREL After Single Shot Injection Ropivacaine Interscalene Nerve Block
Brief Title: Effective Pain Management During Shoulder Replacement Surgery With EXPAREL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-025
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative; Shoulder Osteoarthritis
Keywords: pain control; EXPAREL; shoulder surgery; continuous interscalene nerve block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPAREL (Experimental): Those patients randomized to receive LIA of EXPAREL will have 266mg EXPAREL diluted to 100mL, and drawn into (5) 20mL syringes affixed with (5) 22-gauge needles. Investigators will administer the syringes to the tissue in small increments with the plunger held steady while withdrawn from the tissue to avoid saturating the area around the needle sticks since EXPAREL doesn't readily travel through the tissue.
  Interventions: Drug: local infiltration of liposomal bupivacaine
- interscalene nerve block (Active Comparator): Patients will then receive 0.2% preservative-free ropivacaine at 8mL/hr beginning at the conclusion of surgery and delivered for approximately 50 hours (or finish of 400mL) via elastomeric infusion system (OnQ Pain Relief System: Select A Flow, Kimberly-Clark Corporation, Roswell, Georgia). Patients are instructed prior to discharge how to pull the catheters at home. Patients may also return to surgeon's office for catheter removal once the pain ball is empty if they prefer.
  Interventions: Other: continuous infusion of ropivacaine interscalene nerve block

INTERVENTIONS:
Drug: local infiltration of liposomal bupivacaine — Those patients randomized to receive LIA of EXPAREL will have 266mg EXPAREL diluted to 100mL, and drawn into (5) 20mL syringes affixed with (5) 22-gauge needles. Investigators will administer the syringes to the tissue in small increments with the plunger held steady while withdrawn from the tissue to avoid saturating the area around the needle sticks since EXPAREL doesn't readily travel through the tissue.
  Arms: EXPAREL
Other: continuous infusion of ropivacaine interscalene nerve block — All patients will receive a single injection of 30mL, 0.5% preservative-free ropivacaine.
  Those patients randomized to receive CINB will then have an indwelling catheter placed and held in place by Dermabond and Tegaderm. Placement will be confirmed by ultrasound. Patients will then receive 0.2% preservative-free ropivacaine at 8mL/hr beginning at the conclusion of surgery and delivered for approximately 50 hours (or finish of 400mL) via elastomeric infusion system (OnQ Pain Relief System: Select A Flow, Kimberly-Clark Corporation, Roswell, Georgia). Patients are instructed prior to discharge how to pull the catheters at home. Patients may also return to surgeon's office for catheter removal once the pain ball is empty if they prefer.
  Arms: interscalene nerve block

SUMMARY:
The purpose of this study is to examine the effectiveness of post-operative pain control of local infiltration (LIA) of EXPAREL administration to ropivacaine administered via continuous interscalene nerve block (CINB) for postoperative pain relief following shoulder replacement. Effectiveness will be measured in opioid consumption and NRS pain intensity scores from 0-4h, 4-8h, 9-12h, 13-16h, 17-20, 21-24h, 48 hours and 72 hours post-op. Patient satisfaction with pain control; patient functional outcome; adverse events related to CINB, EXPAREL administration, and opioid consumption; and pain intensity scores from the time of surgery until post-operative day 10 (+/- 5 days) will also be examined.

DETAILED DESCRIPTION:
Shoulder replacement surgery is recognized as having the potential to cause a considerable amount of pain that may require opioid consumption for several days post-operatively. The side effects of opioids are numerous, and ropivacaine administered pre-operatively via interscalene nerve block, with a post-operative continuous ropivacaine infusion through an indwelling catheter (CINB) is a highly effective method for controlling pain and reducing opioid consumption and side effects. While CINB provides adequate post-operative analgesia, and may extend post-operative pain relief for up to 48 hours, there are some risks associated with CINB ranging from catheter tip withdrawal to more serious complications including catheter tip beakage, brachial plexus injury, and pulmonary complications. Local infiltration of liposomal bupivacaine (EXPAREL Pacira Pharmaceuticals, Inc., Parsippany, New Jersey) may provide longer-lasting pain relief when compared to single shot INB (SSINB), and reduce opioid consumption at 24 hours, 48 hours and 72 hours post-op. Studies have shown inconsistency in the effectiveness of EXPAREL, and one proposed reason is the method of administration. Clinicians experienced in their infiltration technique demonstrated greater improvement in pain-related outcomes. The first 48 hours post-op present the most likely opportunity for reducing narcotic administration, which increases the value of attempting to reduce opioid consumption during this period. The cost of EXPAREL LIA, is slightly less than the cost of CINB, and if pain control is comparable, may benefit the patient in reducing hospital costs. The purpose of this study is to examine the effectiveness of pain control of local infiltration of EXPAREL administration to ropivacaine administered via continuous interscalene nerve block (CINB) for postoperative pain relief following shoulder replacement. Effectiveness will be measured in opioid consumption and NRS pain intensity scores from 0-4h, 4-8h, 9-12h, 13-16h, 17-20, 21-24h, 48 hours and 72 hours post-op. Patient satisfaction with pain control; patient functional outcome; adverse events related to CINB, EXPAREL administration, and opioid consumption; and pain intensity scores from the time of surgery until post-operative day 10 (+/- 5 days) will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for primary total shoulder replacement or reverse total shoulder replacement
* Patient must be 18 years or older
* Patient must be willing and able to sign IRB approved informed consent form, and must be able to understand and agree to follow study protocol.

Exclusion Criteria:

* Severe bronchopulmonary disease
* Oxygen dependent
* Existing nerve injury
* BMI > 40
* Coagulation disorders
* Allergy to ropivicaine or bupivacaine
* History of drug or alcohol abuse
* Opioid use within 3 days prior to surgery
* ASA physical status > lll
* Discharge plan to Skilled nursing facility
* Pregnant women
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | post-operative day 1
  Opioid consumption in morphine equivalents within the first 24 hours post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samarian Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers. De-identified results will be shared via publication, and conference.

REFERENCES:
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Borgeat A, Tewes E, Biasca N, Gerber C. Patient-controlled interscalene analgesia with ropivacaine after major shoulder surgery: PCIA vs PCA. Br J Anaesth. 1998 Oct;81(4):603-5. doi: 10.1093/bja/81.4.603. PMID 9924240
- [Background] Ilfeld BM, Morey TE, Enneking FK. Continuous infraclavicular brachial plexus block for postoperative pain control at home: a randomized, double-blinded, placebo-controlled study. Anesthesiology. 2002 Jun;96(6):1297-304. doi: 10.1097/00000542-200206000-00006. PMID 12170039
- [Background] Bjornholdt KT, Jensen JM, Bendtsen TF, Soballe K, Nikolajsen L. Local infiltration analgesia versus continuous interscalene brachial plexus block for shoulder replacement pain: a randomized clinical trial. Eur J Orthop Surg Traumatol. 2015 Dec;25(8):1245-52. doi: 10.1007/s00590-015-1678-2. Epub 2015 Aug 15. PMID 26276164
- [Background] Okoroha KR, Lynch JR, Keller RA, Korona J, Amato C, Rill B, Kolowich PA, Muh SJ. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: a prospective randomized trial. J Shoulder Elbow Surg. 2016 Nov;25(11):1742-1748. doi: 10.1016/j.jse.2016.05.007. Epub 2016 Jul 14. PMID 27422692
- [Background] Hannan CV, Albrecht MJ, Petersen SA, Srikumaran U. Liposomal Bupivacaine vs Interscalene Nerve Block for Pain Control After Shoulder Arthroplasty: A Retrospective Cohort Analysis. Am J Orthop (Belle Mead NJ). 2016 Nov/Dec;45(7):424-430. PMID 28005096
- [Background] Jefferey D. Angel M, Chris A. Steel JR, Devin Ong, PhD, Heather Watson, PhD, Scott T. Lovald, PhD. Pain Control after Total and Reverse Shoulder Arthroplasty: Interscalene Block vs. Liposomal Bupivacaine. In: AAOS Annual Meeting. 2016
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178